CLINICAL TRIAL: NCT01220297
Title: Sirolimus and Mycophenolate Mofetil as GvHD Prophylaxis in Myeloablative, Matched Related Donor Hematopoietic Cell Transplantation
Brief Title: Sirolimus & Mycophenolate Mofetil as GvHD Prophylaxis in Myeloablative, Matched Related Donor HCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Laura Johnston, Associate Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-14913; SU-09092009-3841 (Other: Stanford University); BMT209 (Other: OnCore)
Record Dates: First submitted 2009-11-24; First posted 2010-10-13 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Hematologic Diseases; Acute-graft-versus-host Disease; Leukemia; Non-Hodgkin Lymphoma (NHL); Hodgkin Lymphoma
MeSH Terms: conditions — Hematologic Diseases; Leukemia; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Sirolimus; Mycophenolic Acid; Carmustine; Etoposide; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carmustine Etoposide Cyclophosphamide (Experimental): Carmustine + Etoposide + Cyclophosphamide followed by Sirolimus and Mycophenolate mofetil (MMF) as prophylaxis.
  Interventions: Drug: Sirolimus; Drug: Mycophenolate mofetil (MMF); Drug: Carmustine; Drug: Etoposide; Drug: Cyclophosphamide (Cyclo, CY)
- FTBI + Cyclophosphamide (Experimental): FTBI + Cyclophosphamide followed by Sirolimus and Mycophenolate mofetil (MMF) as prophylaxis.
  Interventions: Drug: Sirolimus; Drug: Mycophenolate mofetil (MMF); Drug: Cyclophosphamide (Cyclo, CY); Drug: FTBI

INTERVENTIONS:
Drug: Sirolimus — Immunosuppressant administered orally to:
  * Adults (age 14 and older), beginning on Day -3 with 12 mg loading dose, followed by 4 mg/day.
  * Children < 13 years or weighing 40 kg, beginning on Day -3 with 3 mg/m² loading dose, followed by 1 mg/ m², rounded to the nearest full milligram.
  Daily dosage may be adjusted to maintain a target serum trough level of 3 to 12 ng/ml. Sirolimus dose tapering will begin at Day 100 in the absence of GvHD, with the goal of discontinuation by 6 months.
  Other Names: Rapamycin; Rapamune
Drug: Mycophenolate mofetil (MMF) — Immunosuppressant given intravenously (IV) at 15 mg/kg 3 times daily, starting on Day 0 ≥ 2 hr after the completion of the HSCT infusion. Dose of MMF will be based on actual body weight, but limited to 15 kg above ideal body weight. MMF dose tapering will begin at Day 100 in the absence of GvHD, with the goal of discontinuation by 6 months.
  Other Names: Cellcept
Drug: Carmustine — For Carmustine + Etoposide + Cyclophosphamide cohort, chemotherapy administered IV on Day -6 at the lesser of 15 mg/kg or 550 mg/m².
  Other Names: Bis-chloroethylnitrosourea (BCNU, BiCNU)
  Arms: Carmustine Etoposide Cyclophosphamide
Drug: Etoposide — For Carmustine + Etoposide + Cyclophosphamide cohort, chemotherapy administered IV on Day -4 at 60 mg/kg
  Other Names: VP-16; VP16
  Arms: Carmustine Etoposide Cyclophosphamide
Drug: Cyclophosphamide (Cyclo, CY) — Cyclophosphamide is a chemotherapy agent.
  For FTBI + Cyclophosphamide cohort, administered IV on Day -3 and -2 at 60 mg/kg.
  For Carmustine + Etoposide + Cyclophosphamide cohort, administered IV on Day -2 at 100 mg/kg
  Other Names: Cytophosphane; Endoxan
Drug: FTBI — For FTBI + Cyclophosphamide cohort, administered as 1320 cGy delivered in 11 120 cGy fractions over 4 days starting on Day -7.
  Other Names: total body irradiation
  Arms: FTBI + Cyclophosphamide

SUMMARY:
A continuation study of sirolimus and mycophenolate mofetil (MMF) for graft-vs-host disease (GvHD) prophylaxis for patients undergoing matched related allogeneic hematopoietic stem cell transplantation (HSCT) for acute and chronic leukemia, myelodysplastic syndrome (MDS), high risk non-Hodgkin lymphoma (NHL), or Hodgkin lymphoma (HL)

DETAILED DESCRIPTION:
To explore the novel combination of sirolimus and mycophenolate mofetil (MMF) as graft-vs-host disease (GvHD) prevention in human leukocyte antigen (HLA)-matched related donor peripheral blood stem cell (PBSC) or marrow transplantation (BMT), collectively hematopoietic stem cell transplantation (HSCT). This study will report the toxicities associated with this drug combination.

For all treatments and procedures, Study Day is based on the day of HSCT as Day 0.

ELIGIBILITY:
INCLUSION CRITERIA

* Acute myelogenous leukemia (AML), beyond 2nd remission or relapsed/refractory disease, age 2 to 60 years
* AML, in first or subsequent remission or relapsed/refractory disease, age 51 to 60 years of age
* AML with multilineage dysplasia
* Acute lymphoblastic leukemia (ALL), beyond 2nd remission or relapsed/refractory disease, age 2 to 60 years
* ALL, age 51 - 60 years in first or subsequent remission or relapsed/refractory disease
* Chronic myeloid leukemia (CML), beyond 2nd chronic phase or in blast crisis
* Myelodysplastic syndrome (MDS), including World Health Organization (WHO)classifications of refractory anemia with excess blasts-1 (RAEB-1), RAEB-2 and therapy-related MDS
* MDS with poor long-term survival including myeloid metaplasia and myelofibrosis
* Myeloproliferative disorders
* High-risk non-Hodgkin lymphoma (NHL) in 1st emission
* Relapsed or refractory NHL
* Hodgkin lymphoma (HL) beyond first remission
* Males and females of any ethnic background, 2 to 60 years of age
* Karnofsky Performance Status (KPS) ≥ 70% or Lansky performance status > 70% for patients < 16 years of age.
* Related, matched-donor identified [6/6 human leukocyte antigen (HLA)-A, B and DRB1]
* Willingness to take oral medications during the transplantation period
* Ability to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA

* Prior myeloablative allogeneic or autologous hematopoietic stem cell transplant (HSCT)
* HIV infection
* Pregnant
* Lactating
* Evidence of uncontrolled active infection
* Serum creatinine > 1.5 mg/dL or 24-hour creatinine clearance < 50 mL/min
* Direct bilirubin, Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 x upper limit of normal (ULN)
* Carbon monoxide diffusing capacity (DlCO) < 60% predicted (adults) OR and in-room air oxygen saturation < 92% (children)
* Left ventricular ejection fraction < 45% (adults) OR shortening fraction < 26%(children)
* Fasting cholesterol > 300 mg/dL or Triglycerides > 300 mg/dL while on lipid-lowering agents.
* Receiving investigational drugs unless cleared by the Principal Investigator (PI).
* Prior malignancies except basal cell carcinoma or treated carcinoma in-situ.
* Cancer treated with curative intent ≤ 5 years (EXCEPTION BY PI DISCRETION) (Cancer treated with curative intent > 5 years will be allowed).

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2006-08; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnston, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Graft-vs-Host Disease (GvHD) Prophlyaxis: Sirolimus & Mycophenolate Mofetil as GvHD Prophylaxis in Myeloablative
Period: Overall Study
Arm/Group | Graft-vs-Host Disease (GvHD) Prophlyaxis
Started | 3
Completed | 0
Not Completed | 3
Not completed — Death | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo: Graft-vs-host disease (GvHD) prophylaxis of sirolimus & mycophenolate mofetil (MMF) after chemotherapeutic regimen of carmustine (BCNU) + etoposide (VP-16) + cyclophosphamide (Cyclo)
- GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo: Graft-vs-host disease (GvHD) prophylaxis of sirolimus & mycophenolate mofetil (MMF) after therapeutic regimen of cyclophosphamide (Cyclo) chemotherapy and fractionated total body irradiation (FTBI)
- Total: Total of all reporting groups
Arm/Group | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo | Total
Number analyzed (Participants) | 0 | 3 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 3 | 3
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 1
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 1 | 1
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 2 | 2
Disease Characteristics [Count of Participants; unit: Participants]
  Acute Lymphoblastic Leukemia (ALL) |  | 1 | 1
  Acute Myeloid Leukemia (AML) |  | 1 | 1
  Biphenotypic Acute Leukaemia (BAL) |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Acute Graft-vs-Host Disease (GvHD) (Grade 2 to 4)
Description: Assessed as the incidence of grade 2 to 4 acute graft-vs-host disease (GvHD) at Day 100 post-transplant.
  Stage of Acute GvHD was assessed as follows.
  * Stage 1: Skin: rash < 25% of skin. Liver: bilirubin 2 to 3 mg/dL. Gut: diarrhea > 500 mL/day or persistent nausea with positive biopsy for GvHD
  * Stage 2: Skin: rash 25 to 50% of skin. Liver: bilirubin 3 to 6 mg/dL. Gut: diarrhea >1000 mL/day.
  * Stage 3: Skin: rash > 50% of skin. Liver: bilirubin 6 to 15 mg/dL. Gut: diarrhea > 1500 mL/day.
  * Stage 4: Skin: generalized erythroderma with bulla formation. Liver: bilirubin > 15 mg/dL. Gut: severe abdominal pain with or without ileus
  Grade of Acute GvHD was determined as follows.
  * Grade 1: Stage 1-2 Skin + No Liver stage + No Gut stage
  * Grade 2: Stage 3 Skin OR Stage 1 Liver or Stage 1 Gut
  * Grade 3: No Skin stage + Stage 2 to 3 Liver Stage 2 to 4 Gut
  * Grade 4: Stage 4 Skin + or Stage 2 to 3 Liver + No Gut stage
Time Frame: 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo
Number analyzed (Participants) | 0 | 3
Participants | 0 | 1

2. Secondary Outcome: Acute GvHD (Grade 3 to 4)
Description: Assessed as the incidence of grade 3 to 4 acute GvHD at Day 100 post-transplant.
  Stage of Acute GvHD was assessed as follows.
  * Stage 1: Skin: rash < 25% of skin. Liver: bilirubin 2 to 3 mg/dL. Gut: diarrhea > 500 mL/day or persistent nausea with positive biopsy for GvHD
  * Stage 2: Skin: rash 25 to 50% of skin. Liver: bilirubin 3 to 6 mg/dL. Gut: diarrhea >1000 mL/day.
  * Stage 3: Skin: rash > 50% of skin. Liver: bilirubin 6 to 15 mg/dL. Gut: diarrhea > 1500 mL/day.
  * Stage 4: Skin: generalized erythroderma with bulla formation. Liver: bilirubin > 15 mg/dL. Gut: severe abdominal pain with or without ileus
  Grade of Acute GvHD was determined as follows.
  * Grade 1: Stage 1-2 Skin + No Liver stage + No Gut stage
  * Grade 2: Stage 3 Skin OR Stage 1 Liver or Stage 1 Gut
  * Grade 3: No Skin stage + Stage 2 to 3 Liver Stage 2 to 4 Gut
  * Grade 4: Stage 4 Skin + or Stage 2 to 3 Liver + No Gut stage
Time Frame: 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo
Number analyzed (Participants) | 0 | 3
Participants | 0 | 1

3. Secondary Outcome: Disease-free Survival (DFS)
Description: Assessed as survival without recurrence of disease
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo
Number analyzed (Participants) | 0 | 3
Participants | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from enrollment to time of death or last follow-up, within 2 years.
Time Frame: 2 years
Measure: Median (Full Range); unit: Days
Arm/Group | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo
Number analyzed (Participants) | 0 | 3
Days |  | 405 [72 to 423]

5. Secondary Outcome: Veno-occlusive Disease (VoD)
Description: Assessed as the incidence of veno-occlusive disease (VoD) at 100 days post-transplant.
Time Frame: 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo
Number analyzed (Participants) | 0 | 3
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo
All-Cause Mortality (participants affected / at risk) | 0/0 | 3/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 3/3
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo (N=0) | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo (N=3)
Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Lung (pneumonia)
Veno-occlusive disease (VOD) (Renal and urinary disorders) | 0 (0) | 1 (1) — Hepatobiliary/pancreas
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (3) — including gross hematuria and/or clotted blood in urine
Fever (General disorders) | 0 (0) | 1 (1)
Neutropenic fever (Infections and infestations) | 0 (0) | 2 (3)
AML relapsed (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Centrilobular nodularity (Cardiac disorders) | 0 (0) | 1 (1)
Macular erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Macular erythema on chest/torso/shoulders (darkening confluent) with hyperpigmented macular rash on > 50% body surface area (BSA).
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — dry cough with intermittent sputum production
Acute graft vs host disease (GvHD) (Infections and infestations) | 0 (0) | 2 (2) — Acute GvHD, with skin rash to trunk, upper back, pruritic at times
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — lung infection
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — Due to Pseudomonas bacteremia
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urgency to urinate (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesicles (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Bullae on right arm and torso
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GvHD Prophylaxis of Sirolimus & MMF After BCNU+VP16+Cyclo (N=0) | GvHD Prophylaxis of Sirolimus & MMF After FTBI + Cyclo (N=3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal cramping (Gastrointestinal disorders) | 0 (0) | 2 (2) — Including: Pain, swelling
BLE Numbness (General disorders) | 0 (0) | 1 (2)
Congestion, Nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dehydration (General disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (General disorders) | 0 (0) | 3 (4) — include: light headedness
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — includes: limbs
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hallucinations (General disorders) | 0 (0) | 1 (1)
Hand Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — including: tremors
Headaches (General disorders) | 0 (0) | 1 (1)
Hemorrhoidal Pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypoxia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Klebsiella pneumoniae (Infections and infestations) | 0 (0) | 1 (1) — Infection
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (8)
Neuropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Pressure ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — (orthostatic hypotension)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Thrush (Infections and infestations) | 0 (0) | 2 (2)
Toe pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Weakness (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Rigoring (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Multifocal Pneumonia (Infections and infestations) | 0 (0) | 0 (0)
Madibular pain (General disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No